CLINICAL TRIAL: NCT04925414
Title: Migraine and High Flow Oxygenotherapy at the Emergency Department
Brief Title: Migraine and High Flow Oxygenotherapy at the Emergency Department (MiOx)
Acronym: MiOx
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Nice (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 20-AOI-08
Record Dates: First submitted 2021-05-17; First posted 2021-06-14 (Actual); Last update posted 2024-11-18 (Actual); Status verified 2024-11

CONDITIONS: Migraine
MeSH Terms: conditions — Migraine Disorders

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- oxygenotherapy (Experimental)
  Interventions: Drug: oxygenotherapy
- placebo air aerosol (Placebo Comparator)
  Interventions: Drug: placebo air aerosol

INTERVENTIONS:
Drug: oxygenotherapy — High concentration mask delivering 15L/min of oxygen
  Arms: oxygenotherapy
Drug: placebo air aerosol — High concentration mask delivering 15L/min of air
  Arms: placebo air aerosol

SUMMARY:
Migraine is a common pathology, affecting around 12% of the general population, up to 25% in some cohorts, as well as a significant part of the reasons for emergency room visits.

Unlike cluster headaches, the use of high-flow oxygen therapy has not yet been validated in patients with migraine.

However, several aspects of its pathophysiology, still studied to this day, suggest that the use of normobaric oxygen could have beneficial effects on migraine attacks: tissue hypoxia, cerebrovascular dysfunction with vasodilation, inflammation, etc.

In addition, high-flow oxygen therapy has no significant side effects and almost no contraindication (mainly COPD and other chronic respiratory failure) Its use in the event of a migraine attack would thus allow less recourse to conventional analgesics (with significant side effects for some), a shorter stay in the emergency room, and therefore a benefit in terms of cost and relief for the patient.

In this context, the sponsor wish to carry out a multicenter prospective interventional, single-blind randomized placebo-controlled in parallel groups study.

DETAILED DESCRIPTION:
Migraine is a common pathology, affecting around 12% of the general population, up to 25% in some cohorts, as well as a significant part of the reasons for emergency room visits.

Unlike cluster headaches, the use of high-flow oxygen therapy has not yet been validated in patients with migraine.

However, several aspects of its pathophysiology, still studied to this day, suggest that the use of normobaric oxygen could have beneficial effects on migraine attacks: tissue hypoxia, cerebrovascular dysfunction with vasodilation, inflammation, etc.

In addition, high-flow oxygen therapy has no significant side effects and almost no contraindication (mainly COPD and other chronic respiratory failure) Its use in the event of a migraine attack would thus allow less recourse to conventional analgesics (with significant side effects for some), a shorter stay in the emergency room, and therefore a benefit in terms of cost and relief for the patient.

In this context, the sponsor wish to carry out a multicenter prospective interventional, single-blind randomized placebo-controlled in parallel groups study.

ELIGIBILITY:
Inclusion Criteria:

* 18 years old or more
* Affiliated to a french public health insurance
* ED admission for migraine evocative headache, regarding ICHD3 criterions
* written informed consent

Exclusion Criteria:

* COPD or other chronic respiratory failure conditions
* Pregnant or breastfeeding women or women of childbearing potential not using any means of contraception. A pregnancy test will be performed for women of childbearing age. The results will be communicated to the patient by a doctor of her choice.
* Under legal protection
* Patients who have received treatment with triptan in the past 2 weeks
* Patients who have consumed NSAIDs in the hour before the doctor's examination
* State of migraine headache (crippling attack for more than 72 hours)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2023-10-01 (Actual); Primary Completion 2025-04 (Estimated); Study Completion 2025-04 (Estimated)

PRIMARY OUTCOMES:
Pain evaluation | 30 minutes after aerosol started
  Simple 0-10 pain verbal numerical rating scale (0 being the minimum : no pain, and 10 the maximum : worst pain imaginable by the subject)

SECONDARY OUTCOMES:
Associated symptoms resolution | From aerosol start to 90 minutes after
  Associated symptoms (nausea, photophoby, neurological troubles ) resolution
Assess pain level | From 30 minutes after aerosol start to 90 minutes after
  Simple 0-10 pain verbal numerical rating scale
Occurrence of side effects | From aerosol start to ED exit assesed up to 6 hours, an average of 3 hours
  Evaluate the occurrence of side effects
Assessing time spent in emergencies | From ED admission to exit or transfert assesed up to 6 hours, an average of 3 hours
  Patient stay in the ED duration
Rescue analgesics usage | From ED admission to exit or transfert assesed up to 6 hours, an average of 3 hours
  The frequency of analgesics administration during patients stay

CONTACTS AND LOCATIONS:
Locations (1):
- CHU de Nice, Nice, France

IPD SHARING:
Plan to Share IPD: No
No data sharing is planned